CLINICAL TRIAL: NCT02284373
Title: Randomized Clinical Trial of Pneumatic Compression Device for the Treatment of Venous Ulcers and Lymphedema
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-01568
Record Dates: First submitted 2014-10-22; First posted 2014-11-06 (Estimated); Results first posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Intervention Model Description: This investigation is a randomized clinical trial of a prospective cohort of subjects with venous ulcers, with an observational cohort of 50 subjects with lymphedema. Venous ulcer subjects will be randomized into two arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Randomization Arm 1: (Other): 70 subjects with venous ulcers will receive pneumatic compression with the Flexitouch® for the duration of one month in addition to routine care of venous ulcers and lymphedema. A pre- and post-PCD treatment CIVIQ-2 quality of life questionnaire will be administered to the subjects. For subjects with venous ulcers, wound area pre- and post-treatment will be recorded
  Interventions: Other: Flexitouch for 1 month in addition to routine wound care
- Randomization Arm 2: (Other): 70 subjects with venous ulcers will receive routine care of venous ulcers and lymphedema. A quality of life questionnaire will be administered at enrollment and again after one month. For subjects with venous ulcers, wound area pre- and post-treatment will be recorded.
  Interventions: Other: Routine wound care for venous ulcers and lymphedema
- Observational Arm 3 (Other): 50 subjects with lymphedema will ALL receive PCD treatment. A pre-and post- PCD treatment CIVIQ-2 QOL questionnaire will be administered to all subjects at enrollment and again after one month of treatment.
  Interventions: Device: Flexitouch pneumonic compression

INTERVENTIONS:
Other: Flexitouch for 1 month in addition to routine wound care — simultaneous wound care and pneumonic compression
  Arms: Randomization Arm 1:
Other: Routine wound care for venous ulcers and lymphedema — wound care /dressings
  Arms: Randomization Arm 2:
Device: Flexitouch pneumonic compression — pneumonic compression only
  Arms: Observational Arm 3

SUMMARY:
The purpose of this study is to evaluate the effect of pneumatic compression in improving symptoms, quality of life and wound healing in patients with venous ulcers and/or lymphedema.

DETAILED DESCRIPTION:
This investigation is a randomized clinical trial of a prospective cohort of an estimated 140 subjects with venous ulcers, with an observational cohort of 50 subjects with lymphedema. Venous ulcer subjects will be randomized into two arms:

Randomization Arm 1: 70 subjects with venous ulcers will receive pneumatic compression with the Flexitouch® for the duration of one month in addition to routine care of venous ulcers and lymphedema. A pre- and post-PCD treatment CIVIQ-2 quality of life questionnaire will be administered to the subjects. For subjects with venous ulcers, wound area pre- and post-treatment will be recorded.

Randomization Arm 2: 70 subjects with venous ulcers will receive routine care of venous ulcers and lymphedema. A quality of life questionnaire will be administered at enrollment and again after one month. For subjects with venous ulcers, wound area pre- and post-treatment will be recorded.

Observational Arm 3: 50 subjects with lymphedema will ALL receive PCD treatment. A pre-and post- PCD treatment CIVIQ-2 QOL questionnaire will be administered to all subjects at enrollment and again after one month of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a venous ulcer on the lower extremity for at least 12 weeks14 days
* Presence of lymphedema in the lower extremity for at least 14 days

Exclusion Criteria:

* Pregnant women or women of childbearing potential not on contraception
* Previous use of the pneumatic compression device
* Class IV congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-05; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Randomization Arm 1: | Randomization Arm 2: | Observational Arm 3
Started | 5 | 5 | 29
Completed | 5 | 2 | 29
Not Completed | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Other | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomization Arm 1: | Randomization Arm 2: | Observational Arm 3 | Total
Number analyzed (Participants) | 5 | 2 | 29 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 12 | 14
  >=65 years | 4 | 1 | 17 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 14 | 18
  Male | 2 | 1 | 15 | 18
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 29 | 36

OUTCOME MEASURES:

1. Primary Outcome: To Assess Quality of Life in Patients With Lymphedema and Venous Ulcers Using CIVIQ-2 Self Questionnaire
Description: Study was terminated due to inadequate enrollment. No data was collected for this outcome measure.
Time Frame: 30 days
Population: Study was terminated due to inadequate enrollment. No data was collected for this outcome measure.
Arm/Group | Randomization Arm 1: | Randomization Arm 2: | Observational Arm 3
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | Randomization Arm 1: | Randomization Arm 2: | Observational Arm 3
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/2 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2 | 0/29
Other Adverse Events (participants affected / at risk) | 0/5 | 0/2 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No